CLINICAL TRIAL: NCT06865313
Title: Total or Subtotal Maxillectomy with Scapular Free Flap Reconstruction: Airway Management, Aesthetic and Functional Results
Brief Title: Functional Evaluation After Maxillectomy and Scapular Free Flap Reconstruction
Status: Completed | Type: Observational
Sponsor: Hôpital de la Croix-Rousse (Other)
Responsible Party: Principal Investigator, SAYAH Charline, Doctor, Hôpital de la Croix-Rousse
Other Study IDs: 2023-05-022-CS
Record Dates: First submitted 2025-02-18; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Maxillary Sinus Squamous Cell Carcinoma
Keywords: Maxillectomy; Reconstruction; Scapula; Tracheotomy; Functional; Aesthetic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients studied: patients with malignant or benign maxillary sinus tumors managed by total maxillectomy and free scapular flap reconstruction

SUMMARY:
The goal of the study is to analyse the functional and aesthetic outcomes after removal of the maxillar bone and reconstruction with part of the scapular bone for people having maxillary tumor

ELIGIBILITY:
Inclusion Criteria:

* Patient with maxillary sinus tumor
* Treated by maxillectomy with free scapula tip flap reconstruction
* 18 years of age or older

Exclusion Criteria:

* Reconstruction failure
* Carcinomatous recurrence and/or further progression impacting quality of life
* Death

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients with malignant or benign maxillary sinus tumors managed by total maxillectomy and free scapula tip flap reconstruction between January 2015 and July 2023 in the Ear-Nose-Throat (ENT) department of Croix Rousse Hospital in Lyon, France.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
time to resumption of oral feeding | through study completion, an average of 15 days
  time to resumption of oral feeding after the surgery, measuring in days
duration of hospitalization in a continuing care unit | through study completion, an average of 15 days
  hospitalization in a continuing care unit after the surgery, measuring in days
Tracheotomy | through study completion, an average of 15 days
  need to do a tracheotomy during or after the surgery, qualitative outcome (yes or no)
Hospitalisation time | through study completion, an average of 15 days
  Duration of the whole hospitalisation in the ENT unit, measuring in days

SECONDARY OUTCOMES:
Swallowing assessment with the Functional Oral Intake Scale | through study completion, an average of 2 years
  Swallowing was assessed using the Functional Oral Intake Scale (FOIS). Scores ranged from one (no oral intake) to seven (normal diet with no change in texture), with a high score indicating good swallowing function.
Aesthetic evaluation | through study completion, an average of 2 years
  A subjective patient assessment of the aesthetic result was carried out using the appearance subcategory of the University of Washington Quality of Life Questionnaire (UW-QOL v4). There are five possible responses, each scored at 0, 25, 50, 75 and 100. A score of 0 represents the worst possible aesthetic result, and a score of 100 the best possible result.
Quality of Life assessment using European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-C30 (version 3.0) and European Organisation for Research and Treatment of Cancer Head & Neck 43 questionnaires. | through study completion, an average of 2 years
  The QLQ-C30 is a general quality-of-life questionnaire specific to oncological pathology and intended for all cancer patients regardless of location.
  It comprises a central questionnaire for assessing 5 functions (physical, cognitive, social, limitations in daily activities and psychological), 9 symptoms and overall health. To this questionnaire can be added modules specific to a cancer site, such as the EORTC QLQ-H&N43 for head and neck cancers.
  Responses to both questionnaires are then transformed to produce a score ranging from 0 to 100. For the functional scales and the global health scale, a high score represents a good level of functioning, while a high score on the symptom scales indicates a high level of symptoms and/or problems.
Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire | through study completion, an average of 2 years
  Functional assessment of the upper limb was performed using the Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire. This is a subjective self-assessment questionnaire of the overall functional capacity of both upper limbs. The score ranges from 0 to 100. Higher scores indicate an inability to perform tasks, great difficulty in doing them, or significant symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Carine FUCHSMANN, Principal Investigator — Hospice Civil de Lyon
Locations (1):
- Croix Rousse Hospital, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided